CLINICAL TRIAL: NCT03809923
Title: Effects of Combination Intravenous Dexmedetomidine and Lidocaine on Postoperative Nausea and Vomiting After Laparoscopic Hysterectomy With General Anesthesia
Brief Title: Dexmedetomidine Combined With Lidocaine Infusion Affect PONV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anqing Municipal Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: xuwen
Record Dates: First submitted 2019-01-16; First posted 2019-01-18 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Lidocaine; Dexmedetomidine; Nausea and Vomiting, Postoperative
Keywords: Lidocaine; Dexmedetomidine; Postoperative nausea and vomiting; laparoscopic hysterectomy
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Lidocaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dexmedetomidine Combined With Lidocaine Infusion Affect PONV (Experimental)
  Interventions: Drug: lidocaine and dexmedetomidine infusion; Drug: Saline infusion; Drug: Lidocaine infusion; Drug: Dexmedetomidine infusion
- Effect of infusion saline on PONV (Experimental)
  Interventions: Drug: lidocaine and dexmedetomidine infusion; Drug: Saline infusion; Drug: Lidocaine infusion; Drug: Dexmedetomidine infusion
- Effect of infusion lidocaine on PONV (Experimental)
  Interventions: Drug: lidocaine and dexmedetomidine infusion; Drug: Saline infusion; Drug: Lidocaine infusion; Drug: Dexmedetomidine infusion
- Effect of infusion dexmedetomidine on PONV (Experimental)
  Interventions: Drug: lidocaine and dexmedetomidine infusion; Drug: Saline infusion; Drug: Lidocaine infusion; Drug: Dexmedetomidine infusion

INTERVENTIONS:
Drug: lidocaine and dexmedetomidine infusion — Patients received IV bolus infusion of lidocaine (2%) 1.5 mg/kg and dexmedetomidine 0.5 µg/kg diluted with normal saline to 20 ml in the LD group respectively, over 10 minutes before induction of anesthesia, followed by a continuous IV infusion at rate of lidocaine 1.5 mg/kg and dexmedetomidine 0.4 µg/kg made up to 20 mL every hour until 30 min before the end of operation, respectively.
Drug: Saline infusion — Patients received 20 ml normal saline and 20 ml normal saline in the CON group respectively, over 10 minutes before induction of anesthesia, followed by a continuous IV infusion 20 ml normal saline and 20 ml normal saline every hour until 30 min before the end of surgery
Drug: Lidocaine infusion — patients received an IV bolus infusion of lidocaine (2%) 1.5 mg/kg made to 20ml with normal saline and 20ml normal saline respectively, over 10 minutes before induction of anesthesia, followed by a continuous IV infusion of lidocaine 1.5 mg/kg made up to 20ml and 20ml normal saline every hour until 30 min before the end of operation, respectively.
Drug: Dexmedetomidine infusion — Patients received IV bolus infusion of dexmedetomidine 0.5 μg/kg made to 20ml with normal saline and 20ml normal saline respectively, over 10 minutes before induction of anesthesia, followed by a continuous IV infusion of dexmedetomidine 0.4μg/kg made up to 20ml and 20ml normal saline every houruntil 30 min before the end of operation, respectively.
  Other Names: Dexmedetomidine

SUMMARY:
BACKGROUND: Few researches have manifested that intravenous (IV) lidocaine or dexmedetomidine decreased the incidence of postoperative nausea and vomiting (PONV). The investigators investigated whether IV lidocaine plus dexmedetomidine infusion could better reduce the incidence of PONV after laparoscopic hysterectomy.

METHODS: Two hundred and forty women with elective laparoscopic hysterectomy were randomly divided into four groups: the control group (group C, n=60) received an equal volume of saline, the lidocaine group (group L, n=60) received IV lidocaine (bolus infusion of 1.5 mg/kg over 10 min, 1.5 mg/kg/h continuous infusion), the dexmedetomidine group (group D, n=60) received dexmedetomidine administration (bolus infusion of 0.5 µg/kg over 10 min, 0.4 µg/kg/h continuous infusion), the lidocaine plus dexmedetomidine group (group LD, n=60) received combination of lidocaine (bolus infusion of 1.5 mg/kg over 10 min, 1.5 mg/kg/h continuous infusion) and dexmedetomidine administration (bolus infusion of 0.5 µg/kg over 10 min, 0.4 µg/kg/h continuous infusion). Primary outcome was the incidence of the first 48 h nausea, vomiting and PONV after surgery. The secondary outcomes included perioperative propofol and remifentanil consumption, postoperative fentanyl requirement, Ramsay sedation score, and bradycardia during post-anaesthesia care unit (PACU) stay.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical statusⅠand Ⅱ
* Aged 40-60 years
* Scheduled for elective laparoscopic hysterectomy

Exclusion Criteria:

* History of allergy to local anesthetics
* BMI>30
* Severe respiratory disease
* Renal or hepatic insufficiency
* History of preoperative opioids medication and psychiatric
* preoperative bradycardia
* preoperative atrioventricular block
* Subjects who experienced severe hypotension (mean arterial pressure [MAP] <60 mmHg) or bradycardia (heart rate [HR] <40 bpm), urticaria, or arrhythmia during lidocaine and dexmedetomidine infusion period

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
postoperative nausea | 0-2 hours after surgery
  Our primary outcome was the incidence of nausea during the 0-2 hours after surgery
postoperative nausea | 2-24 hours after surgery
  Our primary outcome was the incidence of nausea during the 2-24 hours after surgery
postoperative nausea | 24-48 hours after surgery
  Our primary outcome was the incidence of nausea during the 24-48 hours after surgery
postoperative vomiting | 0-2 hours after surgery
  Our primary outcome was the incidence of vomiting during the 0-2 hours after surgery
postoperative vomiting | 2-24 hours after surgery
  Our primary outcome was the incidence of vomiting during the 2-24 hours after surgery
postoperative vomiting | 24-48 hours after surgery
  Our primary outcome was the incidence of vomiting during the 24-48 hours after surgery
postoperative nausea and vomiting (PONV) | 0-2 hours after surgery
  Our primary outcome was the incidence of PONV during the 0-2 hours after surgery
postoperative nausea and vomiting (PONV) | 2-24 hours after surgery
  Our primary outcome was the incidence of PONV during the 2-24 hours after surgery
postoperative nausea and vomiting (PONV) | 24-48 hours after surgery
  Our primary outcome was the incidence of PONV during the 24-48 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anqing Hospital Anesthesiology, Anqing, Anhui, China

REFERENCES:
- [Derived] Xu S, Wang S, Hu S, Ju X, Li Q, Li Y. Effects of lidocaine, dexmedetomidine, and their combination infusion on postoperative nausea and vomiting following laparoscopic hysterectomy: a randomized controlled trial. BMC Anesthesiol. 2021 Aug 4;21(1):199. doi: 10.1186/s12871-021-01420-8. PMID 34348668